CLINICAL TRIAL: NCT02707224
Title: A Randomized, Single-dose, Open, Crossover Clinical Trial to Compare the Pharmacokinetics of DP-R208 (Candesartan Cilexetil and Rosuvastatin Calcium Fixed Dose Combinations) in Comparison to Each Component Administered Alone in Healthy Male Volunteers
Brief Title: Clinical Trial to Compare the Pharmacokinetics of DP-R208
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DP-CTR208-I-02
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: DP-R208
MeSH Terms: interventions — candesartan cilexetil; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): combination dose of Candesartan cilexetil and Rosuvastatin and DP-R208 in order
  Interventions: Drug: DP-R208; Drug: Candesartan cilexetil; Drug: Rosuvastatin
- Group B (Experimental): DP-R208 and combination dose of Candesartan cilexetil and Rosuvastatin in order
  Interventions: Drug: DP-R208; Drug: Candesartan cilexetil; Drug: Rosuvastatin

INTERVENTIONS:
Drug: DP-R208 — Investigational product is prescribed to all of randomized subjects
Drug: Candesartan cilexetil — Investigational product is prescribed to all of randomized subjects
Drug: Rosuvastatin — Investigational product is prescribed to all of randomized subjects

SUMMARY:
A randomized, single-dose, open, crossover clinical trial to compare the pharmacokinetics of DP-R208 (Candesartan cilexetil and Rosuvastatin calcium fixed dose combinations) in comparison to each component administered alone in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* BMI 17.5~30.5
* signed the informed consent form prior to the study participation

Exclusion Criteria:

* Clinically significant disease
* Previously donate whole blood within 60 days or component blood within 14 days
* Clinically significant allergic disease
* Taken IP in other trial within 90 days
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | up to 72 hours post dose
Area under the plasma concentration versus time curve (AUC) | up to 72 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Min-Gul Kim, Ph.D, Principal Investigator — Chonbuk National University Hospital

IPD SHARING:
Plan to Share IPD: No